CLINICAL TRIAL: NCT06050980
Title: A Phase I, Open-label, Dose-escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic of HSK40118 in Patients With EGFR Mutation Locally Advanced or Metastatic NSCLC
Brief Title: Phase I Study of HSK40118 in NSCLC Patients With EGFR Mutation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK40118-101
Record Dates: First submitted 2023-07-17; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase Ia(Part A): HSK40118 as monotherapy (Experimental): Phase 1a(Part A): dose escalation of HSK40118 as monotherapy at various dose levels
  Interventions: Drug: HSK40118
- Phase Ia(Part B): HSK40118 as monotherapy (Experimental): Phase 1a(Part B): dose extention of HSK40118 as monotherapy at certain dose levels
  Interventions: Drug: HSK40118
- Phase Ib: HSK40118 as monotherapy (Experimental): Phase 1b: dose expansion for HSK40118 as monotherapy at a dose determined during Phase 1 in patients with previous treatment with 3rd-generation EGFR-TKI
  Interventions: Drug: HSK40118

INTERVENTIONS:
Drug: HSK40118 — Oral administration, QD

SUMMARY:
This is a phase I, open-label, dose-escalation and expansion study to evaluate the safety, tolerability, PK and PD of HSK40118 when given orally in patients with active EGFR mutation locally advanced or metastatic non-small cell lung cancer (NSCLC).

The study will contain two phase: Phase Ia is dose escalation phase and Phase Ib is dose expansion phase.

DETAILED DESCRIPTION:
Phase Ia will contain two part: Dose Escalation Part(Part A) and Extension Part(Part B). Part A based on the "3+3" design for dose escalation and safety evaluation requirements. Patient cohorts at selected doses may be extended to further investigate the tolerability, PK and PD of HSK40118. The number of patients to be enrolled will be up to 10 subjects in each Part B cohort. Approximately 30-70 subjects will be enrolled in Phase Ia.

Phase Ib no less than 130 subjects will be enrolled in each expansion cohort, cohort A will be enrolled 30-50 subjects, cohort B will be enrolled no less than 100 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, Male and female patients, at time of signing informed consent form (ICF).
2. ECOG=0-1, with no deterioration in 2 weeks before first dose of HSK40118.
3. Histological or cytological confirmed diagnosis of unresectable locally advanced or metastatic NSCLC.
4. Patients will provide blood or tumor sample according to their own willingness.
5. Patients in Phase Ia and Ib will fulfill the different criteria of the following:

   Phase Ia(Part A): Previous treatment with at least one EGFR-TKI, including 1st, 2nd and 3rd-generation EGFR-TKI; Phase Ia(Part B)/Phase Ib: Previous treatment with 3rd-generation EGFR-TKI.
6. tumour lesions/lymph nodes: Phase Ia(Part A): Patients should have at least one assessable tumour lesions/malignant lymph nodes; Phase Ia(Part B) /Phase Ib: Patients should have at least one measurable tumour lesions/malignant lymph nodes.
7. Life expectancy ≥ 3 months.
8. Adequate hematologic and organ function per protocol.
9. Women of childbearing potential (WOCBP) and fertile males with WOCBP partners must use highly effective contraception per protocol throughout and after 90 days of the last dose of the study.

Exclusion Criteria:

1. malignant tumor within 5 years, with the exception of cutaneous squamous cell carcinoma, cervical carcinoma in situ, papillary thyroid carcinoma, or other tumors with low malignancy.
2. Unstable spinal cord compression or brain metastases per protocol.
3. Uncontrollable pleural effusion, ascites, or pericardial effusion per protocol.
4. Prior treatment with 4th-generation EGFR-TKIs(TKI for 3th-generation resistance).
5. Treatment with any of the following:

   Prior treatment with an EGFR-TKI or other small-molecule anti-tumor drug within 7 days or approximately 5 × t1/2 prior to the first dose of HSK40118, whichever is shorter; Prior treatment with chemotherapy, palliative radiotherapy, or Herbal therapy within 2 weeks or approximately 5 × t1/2 prior to the first dose of HSK40118, whichever is shorter; Prior treatment with radiotherapy, immunotherapy/biotherapy therapy, or other pharmaceutical clinical trial within 4 weeks or approximately 5 × t1/2 prior to the first dose of HSK40118, whichever is shorter.
6. Treatment with inhibitors for P-glycoprotein (P-gp) within 7 days prior to the first dose of HSK40118.
7. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment, with the exception of alopecia, dermal toxicity, and other toxicity considering no safety risks by investigator.
8. Any disease which would cause chronic diarrhea, eg. Crohn's disease, or irritable bowel syndrome.
9. Any disease which would preclude drug absorption, metabolism or pharmacokinetics, eg. active peptic ulcer or chronic gastroesophageal reflux disease.
10. Any severe disease of respiratory system, eg. interstitial lung disease, radiation pneumonitis, drug-induced pneumonitis, or uncontrolled asthma.
11. Patient who have clinically significant or uncontrolled cardiac disease, include: QTc interval ≥ 450(male)/470(female) msec; any clinically significant arrhythmia; left ventricular ejection fraction < 50%; myocardial infarction, unstable angina, or class III/IV cardiac failure by the NYHA that occurred within 6 months prior to the first dose of HSK40118.
12. Any thromboembolic events within 6 months prior to the first dose of HSK40118; any familial or aquired thrombophilia.
13. Active bleeding at screening, history of visceral hemorrhage within 3 months prior to the first dose of HSK40118, or visceral bleeding tendency within 6 months prior to the first dose of HSK40118.
14. Patient who is undergoing, or receiving long-term(> 6 months) anticoagulant/antiplatelet therapy; receiving drugs affecting coagulation function 1 week prior to the first dose of HSK40118.
15. INR, APTT > 1.5xULN, or any bleeding tendency or coagulopathy at screening.
16. Uncontroled hypertension(systolic pressure ≥160mmHg, or diastolic pressure ≥100mmHg).
17. Any unstable systemic disease, eg. severe metabolic disease: liver cirrhosis, renal failure, or uremia.
18. Any disease of the eyes > CTCAE v5.0 Grade 1.
19. Autologous transplantation surgery within 3 months prior to the first dose of HSK40118; Allogeneic transplantation, or stem-cell Transplant surgery within 6 months prior to the first dose of HSK40118; Major surgery or significant traumatic injury occurring within 4 weeks prior to the first dose of HSK40118.
20. Patients with HIV, HBV or HCV infection.
21. Patients with active syphilis infection.
22. Patients who have an uncontroled systematic infection, eg. fungal, bacterial, or virus infection.
23. Patients who would interfere with cooperation or outcome-assessment of the trial.
24. Allergic to any HSK40118 active constituent or ingredients.
25. (Child-bearing period women only)Patients testing positive for pregnancy, or during lactation.
26. Any other circumstances that would, in the investigator's judgment, prevent the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2027-06-07 (Estimated)

PRIMARY OUTCOMES:
MTD | Up to approximately 52 months
  MTD determination: dose limiting toxicity (DLT) rate
DLTs | Up to approximately 52 months
  Incidence of dose-limiting toxicities (DLTs) at Cycle 0 and Cycle1
AEs | Up to approximately 52 months
  Rate and severity of adverse events of HSK40118 as monotherapy
Eastern Cooperative Oncology Group Performance Status Scale(ECOG PS) | Up to approximately 52 months
  Change of the grade as a part of HSK40118 safety data. The functional status of patients will be assessed by the ECOG PS, which is described as a scale including grade 0(fully active) to grade 5(dead).

SECONDARY OUTCOMES:
Overall response rate(ORR) | Up to approximately 52 months
  ORR, defined as the proportion of patients who experience a best response of confirmed CR or PR according to RECIST 1.1
Disease control rate (DCR) | Up to approximately 52 months
  DCR, defined as the proportion of patients who experience a best response of CR, PR, or stable disease (SD) according to RECIST 1.1
Duration of response (DOR) | Up to approximately 52 months
  DOR, defined as the time from first documented response of complete response (CR) or partial response (PR) to the date of first documented progressive disease or death due to any cause, whichever occurs first
Progression free survival (PFS) | Up to approximately 52 months
  PFS, defined as the time from the first dose of HSK40118 until the date of first documented progressive disease or death due to any cause, whichever occurs first
Overall survival (OS) | Up to approximately 52 months
  OS, defined as the time from the first dose of HSK40118 until the date of death due to any cause
AUC of HSK40118 | Blood samples will be collected on 6 occasions for each patient throughout study: cycle 0 day 1, cycle 0 day 2, cycle 0 day 3, cycle 1 day 1, cycle 1 day 8 and cycle 1 day 15.
  Pharmacokinetics (PK) parameter of HSK40118. AUC is the definite integral of a curve that describes the variation of a drug concentration in blood plasma as a function of time. AUC reflects the actual body exposure to drug after single dosing and at steady state after multiple dosing.
Cmax of HSK40118 | Blood samples will be collected on 6 occasions for each patient throughout study: cycle 0 day 1, cycle 0 day 2, cycle 0 day 3, cycle 1 day 1, cycle 1 day 8 and cycle 1 day 15.
  Pharmacokinetics (PK) parameter of HSK40118. Cmax is the maximum (or peak) serum concentration that the drug achieves in blood after the drug has been administered.
Cmin of HSK40118 | Blood samples will be collected on 3 occasions for each patient throughout study: cycle 1 day 1, cycle 1 day 8 and cycle 1 day 15.
  Pharmacokinetics (PK) parameter of HSK40118. Cmin is the minimum (or trough) serum concentration that the drug achieves in blood at steady state after multiple dosing.
Tmax of HSK40118 | Blood samples will be collected on 6 occasions for each patient throughout study: cycle 0 day 1, cycle 0 day 2, cycle 0 day 3, cycle 1 day 1, cycle 1 day 8 and cycle 1 day 15.
  Pharmacokinetics (PK) parameter of HSK40118. Tmax is defined as the time of maximum concentration of the drug in blood observed after single dosing and at steady state after multiple dosing.
Terminal half life(t1/2) after single dosing of HSK40118 | Blood samples will be collected on 3 occasions for each patient throughout study: cycle 0 day 1, cycle 0 day 2, cycle 0 day 3.
  Pharmacokinetics (PK) parameter of HSK40118 by assessment of the terminal half-life after single dosing.
CL/F of HSK40118 | Blood samples will be collected on 3 occasions for each patient throughout study: cycle 0 day 1, cycle 0 day 2, cycle 0 day 3.
  Rate and extent of absorption of HSK40118 by assessment of apparent clearance following oral administration.
Vd/F of HSK40118 | Blood samples will be collected on 3 occasions for each patient throughout study: cycle 0 day 1, cycle 0 day 2, cycle 0 day 3.
  Rate and extent of absorption of HSK40118 by assessment of the apprarent volume of distribution.
λz of HSK40118 | Blood samples will be collected on 3 occasions for each patient throughout study: cycle 0 day 1, cycle 0 day 2, cycle 0 day 3.
  Pharmacokinetics (PK) parameter of HSK40118 by assessment of first-order rate constant associated with the terminal (log-linear) portion of the curve.
MRT(Mean residence time) of HSK40118 | Blood samples will be collected on 3 occasions for each patient throughout study: cycle 0 day 1, cycle 0 day 2, cycle 0 day 3.
  Pharmacokinetics (PK) parameter of HSK40118 by assessment of mean residence time, which meas AUMC(Area under the moment curve)/AUC(Area under the curve) of drug concentration in blood plasma.
Cav,ss(average concentration at steady state) of HSK40118 | Blood samples will be collected on 3 occasions for each patient throughout study: cycle 1 day 1, cycle 1 day 8 and cycle 1 day 15.
  Pharmacokinetics (PK) parameter of HSK40118 by assessment of average concentration at steady state after multiple dosing.

OTHER OUTCOMES:
EGFR protein degradation | Tissue samples will be collected on 2 occasions for each patient throughout study: screening period, cycle 1 day 15(±7 days).
  Pharmacodynamics (PD) parameter of HSK40118 by assessment of the percentage of EGFR protein degradation at steady state after multiple dosing.
circulation tumor DNA(ctDNA) | Blood samples will be collected on 3 occasions for each patient throughout study: screening period, cycle 2 day 1, cycle 3 day 1.
  Pharmacodynamics (PD) parameter of HSK40118 by assessment of the concentration of ctDNA after multiple dosing.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Taizhou hospital of Zhejiang Province, Taizhou, Zhejiang